CLINICAL TRIAL: NCT06288061
Title: Effectiveness of Non-invasive Phrenic Nerve Neuromodulation in Subjects With Inflammatory Bowel Disease and Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, María Pérez Montalbán, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Phrenic Nerve Neuromodulation
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases; Neck Pain
MeSH Terms: conditions — Inflammatory Bowel Diseases; Neck Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-invasive Phrenic Nerve Neuromodulation (Experimental)
  Interventions: Device: Non-invasive Neuromodulation
- Cervico-dorsal Massage (Placebo Comparator)
  Interventions: Other: Cervico-dorsal Massage

INTERVENTIONS:
Device: Non-invasive Neuromodulation — This intervention group will receive neuromodulation treatment two days a week for a total of six sessions.
  The patient is placed in the supine position with a cushion under the knees. The physiotherapist will be positioned behind the patient's head on the side to be treated. The technique will be applied on both anterolateral sides of the neck, where the Phrenic nerve passes in front of the anterior Scalene, between the Subclavian arteries and veins. Neuromodulation will be applied with a Pointer Excel II. It will be applied with negative polarity, at a frequency of 2 Hertz (HZ) and with a current intensity varying between 0 and 45 milliamperes (mA). The intensity shall be increased progressively until the patient's diaphragmatic contraction can be observed without pain. The technique shall be applied on each side for a total of 8 minutes, divided into intervals of 10 seconds of stimulation and 20 seconds of rest.
  Arms: Non-invasive Phrenic Nerve Neuromodulation
Other: Cervico-dorsal Massage — This intervention group will receive manual therapy two days a week for a total of six sessions.
  The patient shall be placed prone position with a cushion under his or her feet. This group will receive manual therapy on the entire posterior cervical and dorsal region, the area between the occipital bone, the shoulders and the scapulae. The massage will be carried out with a little oil or cream for about 20 minutes.
  Arms: Cervico-dorsal Massage

SUMMARY:
Inflammatory bowel diseases (IBD) are chronic relapsing diseases that generate an autoimmune response against the bowel and its microbiota. Its prevalence is increasing worldwide. These include Ulcerative Colitis (UC) and Crohn's Disease(CD).

The Phrenic nerve originates at the roots C3-C4-C5 carrying motor and sensory information. Directly or through connections it innervates the diaphragm, pleura, right atrium, pericardium, oesophagus, peritoneum, stomach, falciform and coronary ligaments of the liver, Glisson's capsule, hepatic and inferior vena cava, liver (parenchyma), gallbladder and the rest of the biliary tract, pancreas, small intestine and adrenal glands. It also has fibres of the autonomic nervous system.

Studies show that there is a link between people suffering from IBD and hepatopancreato-biliary diseases. It can therefore generate referred pain to the C3-C4-C5 dermatomes.

Based on the above, the main objective would be to analyse whether non-invasive neuromodulation of the Phrenic nerve reduces neck pain in people with IBD. Secondary objectives were to assess the impact of treatment on quality of life and to study the relationship between IBD and cervical pain.

Hypothesis:

Non-invasive Phrenic nerve neuromodulation in subjects suffering from inflammatory bowel disease and neck pain will improve their quality of live, disability and sensitisation, as well as neck pain and mobility.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's Disease or Ulcerative Colitis.
* Be over 18 years old.
* Disorder of the peridiaphragmatic abdominal viscera.
* Chronic mechanical neck pain.

Exclusion Criteria:

* Previous trauma or surgery to the cervical spine.
* Infection.
* Congenital vertebral anomaly.
* Neurological diseases.
* Signs of neural compression or spinal stenosis.
* Impossibility of applying neuromodulation (fever, pregnancy, pacemaker, epilepsy, neoplastic processes close to the cervical area and skin alterations).
* Severe cognitive impairment and communication deficits.
* Application of physiotherapeutic treatment three months prior to the study.
* Use of analgesics, anti-inflammatory drugs or relaxants in the 24 hours prior to the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
The Visual Analogue Scale (VAS) | The scale shall be measured before starting treatment, before the third session, before the fifth session and two weeks after the last session.
  The Visual Analogue Scale (VAS) consists of a 100 mm line; it indicates the perceived intensity of pain, with zero mm being "no pain" and 100 mm being "the worst pain imaginable".
Cervical mobility | The scale shall be measured before starting treatment, before the third session, before the fifth session and two weeks after the last session.
  It shall be assessed using the iPhone level application. To measure flexion-extension, the mobile will be placed vertically centred on the external auditory canal, obtaining a range of movement between zero and 45-50 degrees. For lateroflexion, it shall be positioned horizontally at the back of the head, giving a range between zero and 45 degrees. For rotations, the mobile shall be positioned vertically on the top of the head, giving a range of movement between zero and 60-80 degrees. Measurements shall be taken with the patient in a seated position. For each movement, three measurements shall be taken to obtain an average value of the three.
The Neck Disability Index (NDI) | The scale shall be measured before starting treatment, before the third session, before the fifth session and two weeks after the last session.
  The Neck Disability Index (NDI) is a questionnaire for the assessment of the functional status of subjects with neck pain. It includes the measurement of 10 items, each scored from zero to five, where zero means "painless" and five means "the most pain imaginable". The points obtained are summed up to obtain a percentage.
The Pressure Pain Threshold (PPT) | The scale shall be measured before starting treatment, before the third session, before the fifth session and two weeks after the last session.
  The Pressure Pain Threshold (PPT) is used to assess pressure pain and is applied with an algometer. The measurement is taken at the medial aspect of the anterior border of the upper trapezius and the spinous process of C4. The assessor shall gradually increase the pressure until the subject indicates with a "yes" when pain or discomfort appears. The patient shall be seated. For each point, three measurements shall be taken to obtain an average value of the three measurements.

SECONDARY OUTCOMES:
The Inflammatory Bowel Disease Questionnaire (IBDQ-32) | The scale shall be measured before starting treatment, before the third session, before the fifth session and two weeks after the last session.
  The Inflammatory Bowel Disease Questionnaire (IBDQ-32) is used to assess health-related quality of life in IBD. The IBDQ-32 questionnaire contains 32 items divided into four items (digestive symptoms, systemic symptoms, emotional and social involvement). Responses are scored from seven to one, with seven being the best score and one being the worst. The total number of points will be added up.
The World Health Organization Quality of Life (WHOQOL-BREF) | The scale shall be measured before starting treatment, before the third session, before the fifth session and two weeks after the last session.
  The World Health Organization Quality of Life (WHOQOL-BREF) is a 26-item scale consisting of four domains (physical health, psychological health, social relationships and environmental health). Each item is scored from one to five, summed to give a score from zero to 100.
The Central Sensitization Inventory (CSI) | The scale shall be measured before starting treatment, before the third session, before the fifth session and two weeks after the last session.
  The Central Sensitisation Inventory (CSI) is a questionnaire to identify patients who have symptoms that may be related to central sensitisation or central sensitisation syndromes. The CSI has two parts, the first includes 25 questions related to common symptoms and the second determines whether the patient has been diagnosed with central sensitisation or related disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Puerto Real, Puerto Real, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Montalban M, Sanchez-Alcala D, Garcia-Dominguez E, Mata-Perdigon FJ, Oliva-Pascual-Vaca A. Effectiveness of Noninvasive Phrenic Nerve Neuromodulation in Subjects With Inflammatory Bowel Disease and Neck Pain: A Randomized Clinical Trial. Neuromodulation. 2025 Oct 30:S1094-7159(25)01036-0. doi: 10.1016/j.neurom.2025.09.311. Online ahead of print. PMID 41171220